CLINICAL TRIAL: NCT01227811
Title: Single Dose, Two-period, Crossover, Fed Bioequivalence Study of Darifenacin Extended Release Oral Formulation (Darisec(R) 15 mg) vs. Enablex(R) 15 mg in Healthy Volunteers.
Brief Title: Single Dose Two-periods Crossover Bioequivalence Study of Darifenacin Tablets in Healthy Volunteers.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Clinical Pharmacology Research Bdbeq S.A. (Other)
Collaborators: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Francisco E. Estevez-Carrizo, M.D. / Principal investigator., Center for Clinical Pharmacology Research Bdbeq S.A.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BDBEQ_DFNLP/ELEA_011
Record Dates: First submitted 2010-10-18; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Bioequivalency
Keywords: Darifenacin; Bioequivalence; Healthy volunteers; Postprandial
MeSH Terms: interventions — darifenacin; Muscarinic Antagonists; Cholinergic Antagonists; Cholinergic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enablex(R) 15 mg , single dose (Active Comparator)
  Interventions: Drug: Darifenacin
- Darifenacin 15 mg tablets, single dose (Experimental)
  Interventions: Drug: Darifenacin

INTERVENTIONS:
Drug: Darifenacin — Single oral dose Darisec(R) 15.0 mg
  Other Names: Muscarinic Antagonists; Cholinergic Antagonists; Cholinergic Agents; Enablex; Darisec
  Arms: Darifenacin 15 mg tablets, single dose
Drug: Darifenacin — Single oral dose Enablex(R) 15 mg
  Arms: Enablex(R) 15 mg , single dose

SUMMARY:
The present study was designed to assess the bioequivalence and pharmacokinetic profiling of a brand generic formulation of darifenacin [Darisec(R)]vs. the innovator [Enablex(R)]in healthy volunteers after a high fat breakfast.

The bioequivalence will be evaluated using:

* the Area Under the Curve (AUC) and,
* the peak plasma concentration (Cmax).

Safety will be evaluated recording:

* vital signs
* adverse events,
* laboratory analysis.
* EKG and chest XRays.

Bioequivalence will be claimed if the drugs comply with local regulatory requirement, eg.:

* mean AUCt/AUCr and 90% confidence interval within 0.80-1.25
* mean Cmaxt/Cmaxr and 90% confidence interval within 0.80-1.25.

DETAILED DESCRIPTION:
Darifenacin is a muscarinic receptor antagonist drug used to treat overactive bladder. There is a new formulation of darifenacin extended release developed by an argentinian pharmaceutical company and, according to regional regulations, a bioequivalence study should be performed to put it in the market.

The purpose of this study is to evaluate the relative bioavailability and pharmacokinetic profiling of a brand generic formulation of darifenacin [Darisec(R) 15 mg] vs. the innovator [Enablex(R) 15 mg] in 24 healthy uruguayan volunteers after a high fat breakfast of 1000 calories (50% fat, 35% carbohydrates (sugar, flour, etc.) and 15& proteins) to establish their average bioequivalence.

The bioequivalence will be evaluated using outcome measures that will be described later.

The pharmacokinetic characteristics of the drugs will be described calculating:

* the time to Cmax (Tmax)
* the elimination constant (Ke),
* the elimination half-life (t1/2e)and,
* the systemic clearance (Cls.

Safety will be evaluated recording:

* vital signs (blood pressure, heart rate, body temperature)
* adverse events,
* laboratory analysis (hemogram, hepatic enzymes, creatinine, sugar in blood,etc.).
* EKG and chest XRays.

Bioequivalence will be claimed if the drugs comply with local and FDA regulatory requirement, eg.:

* mean AUCt/AUCr and 90% confidence interval within 0.80-1.25
* mean Cmaxt/Cmaxr and 90% confidence interval within 0.80-1.25.

Safety will be evaluated comparing incidences of adverse events/adverse effects for both products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 50 years of age (inclusive)
* In good health, as determined by lack of clinically significant abnormalities at screening as judged by the physician.
* Female subjects are required to use a medically accepted method of hormonal contraception or abstinence throughout the entire study period and for one week after the study is completed.
* Body mass index within the range of 18.5 and 29.9 kg/m2 and weight at least 45 kg.

Exclusion Criteria:

* Known hypersensitivity or severe adverse event to darifenacin or similar drugs.
* Urinary retention, narrow-angle glucoma, myasthenia gravis, severe hepatic impairment, severe ulcerative colitis, toxic megacolon.
* Symptomatic hiatus hernia, erosive or symptomatic gastroesophageal reflux disease/heartburn (>2 days in a week), severe constipation, gastrointestinal obstructive disorder, and gastric retention.
* Clinically significant cardiac abnormalities, fainting, low blood pressure upon standing, irregular heartbeats.
* Acute or chronic bronchospastic disease (including asthma and Chronic Obstructive Pulmonary Disease).
* Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis).
* Smokers of more than 5 cigarettes a week.
* Regular use of any drugs known to induce or inhibit hepatic drug metabolism (particularly those that affect CYP2D6) within 30 days prior to each study drug administration.
* Any surgical or medical condition wich might significantly alter the absorption, distribution, metabolism or excretion of drugs which may jeopardize participation in the study.
* Immunodeficiency diseases, including a positive HIV (Elisa or Western blot) test result.
* Positive hepatitis B Surface antigen (HBsAg) or Hepatitis C test result.
* Drug or alcohol abuse within the 6 months prior to dosing.
* Use of prescription drugs within 1 month prior to dosing, or over-the-counter medication (vitamine, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Paracetamol and ibuprofen are acceptable.
* Participation in any clinical investigation within 4 weeks prior to dosing.
* Donation or loss of 400 ml or more of blood within 2 months prior to dosing.
* significant illness within 2 weeks prior to dosing.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Extent of Absorption. | 72 hours
  Extent of absorption will be measured using the area under plasma concentrations of darifenacin vs. time from time 0 to the last sample point (AUC0-t) and from time 0 to infinity (AUC0-inf).
Rate of Absorption | 72
  Rate of abosrption will be measured using the peak concentration of darifenacin (Cmax).

SECONDARY OUTCOMES:
Time to peak concentration (tmax) | 72 hours
  Is the time elapsed from ingestion of darifenacin tablets to plasma peak concentration.
Absorption Rate Constant(Ka) | 72 hours
  The absorption rate constant is the fractional rate of drug disappearance from the intestinal tract, measured in the log-linear phase of drug absorption.
Elimination Rate Constant (Ke) | 72
  The elimiminaiton rate constant is the fractional rate of drug dissapearance from the peripheral compartment, measured in the log-linear phase of elimination.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco E. Estevez-Carrizo, MD, Study Director — Univerisity of Montevideo. Biomedical Science Center.Prudencio de Pena 2440, 11600 Montevideo. Uruguay; Susana Parrillo, M.D., Principal Investigator — Center for Clinical Pharmacology Research Bdbeq S.A., Br. Artigas 1632. c.p. 11600 Montevideo. Uruguay.
Locations (1):
- Center for Clinical Pharmacology Research Bdbeq S.A.; Hospital Italiano de Montevideo.., Montevideo, Montevideo Department, Uruguay

REFERENCES:
- [Background] Skerjanec A. The clinical pharmacokinetics of darifenacin. Clin Pharmacokinet. 2006;45(4):325-50. doi: 10.2165/00003088-200645040-00001. PMID 16584282